CLINICAL TRIAL: NCT06511271
Title: Effect of Progressive Relaxations Applied After Laparoscopic Cholecystectomy on Pain, Nausea and Vomiting
Brief Title: Osmaniye State Hospital"
Acronym: OSH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Osmaniye Korkut Ata University (Other)
Responsible Party: Principal Investigator, Songul Gungor, Phd Lecturer, Osmaniye Korkut Ata University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Osmaniye State Hospital"
Record Dates: First submitted 2024-05-28; First posted 2024-07-19 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: laparoscopic cholecystectomy; Postoperative Pain; nausea; vomiting
MeSH Terms: conditions — Pain, Postoperative; Nausea; Vomiting

STUDY DESIGN:
Intervention Model Description: Patients in the study group underwent progressive relaxation exercises at the 2nd, 6th, 12th and 24th hours after surgery
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (No Intervention): Patients in the control group were given only the standard procedure for laparoscopic cholecystectomy during the research period.
  treatment and care were applied.
- Group 2 (Experimental): The first 10-minute part of the CD audio recordings prepared by the Turkish Psychologists Association is about deep relaxation. purpose; The second 30-minute part includes instructions for relaxation exercises; The last 30 minutes are just It consists of relaxation music[145]. In our study, the instructions in the second part were used. - In addition to standard treatment and care for laparoscopic cholecystectomy, volunteers who accept the study Progressive relaxation exercises were applied by the researcher at the 2nd, 6th, 12th and 24th hours after surgery. When the literature review on PGE was made, it was seen that the application time and frequency of these exercises were not standard; 6th, 12th, 24th hours after surgery; It was applied on the 2nd day after surgery and the total number of sessions varied. It is seen to show. In our study, PGE was detected at the 2nd, 6t
  Interventions: Other: relaxation exercises

INTERVENTIONS:
Other: relaxation exercises — The first 10-minute part of the CD audio recordings prepared by the Turkish Psychologists Association is about deep relaxation.
  purpose; The second 30-minute part includes instructions for relaxation exercises; The last 30 minutes are just consists of relaxation music
  Arms: Group 2

SUMMARY:
Objective: It was conducted as a randomized controlled experimental study to determine the effect of progressive relaxation exercise applied after laparoscopic cholecystectomy on postoperative pain, nausea and vomiting. Method: The population of the study consisted of 105 patients who underwent elective planned laparoscopic cholecystectomy at Osmaniye State Hospital General Surgery Clinic between 25 May and 25 August 2023(Study=38, Control=38). 76 patients, who constituted the sample of the study, were assigned to the study and control groups. Data were collected using the Patient Introduction Form Visual Comparison Scale and Perioperative Patient Monitoring Form.

Patients in the study group underwent progressive relaxation exercises at the 2nd, 6th, 12th and 24th hours after surgery. Frequency, average, Chi-Square test, Independent t-test and Repeated Measures ANOVA test were used to evaluate the data. Results: When the comparison between groups is examined; It was determined that the average pain intensity scores of the patients in the study group at the 6th, 12th and 24th postoperative hours decreased more than the control group and the difference between them was statistically significant (p<0.05). When the comparison between groups is examined; It was determined that the average nausea severity scores of the patients in the study group at the 6th, 12th and 24th postoperative hours decreased significantly compared to the control group and the difference between them was statistically significant (p<0.05). It was determined that there was a decrease in vomiting rates in the study group compared to the control group at the 6th and 12th hours after surgery and the difference between them was significant. Conclusion and Recommendations: It has been determined that progressive relaxation exercises reduces pain, nausea and vomiting after laparoscopic cholecystectomy. In line with the results obtained from the research, it is recommended that nurses teach progressive relaxation exercises to patients and encourage their use, as they are easy to apply to patients and are not an invasive method. Keywords: Laparoscopic cholecystectomy, nausea, nurse, pain, progressive relaxation exercises.

DETAILED DESCRIPTION:
Data were collected at Osmaniye State Hospital General Surgery Clinic between 25 May and 25 August 2023.

Among 76 patients who were hospitalized for laparoscopic cholecystectomy and volunteered to participate in the study (Study group = 38, Control group = 38) was taken. Before starting the application, ;Informed Voluntary ; was obtained from the patients.

Verbal and written permissions were obtained by reading the ; (Annex-I). Working group - Before the patient undergoes surgery, the Patient Information Form (Annex-II) information is obtained from the patient file and asked to the patient.

has been filled.

* The researcher was informed about the surgical intervention, expected nausea and vomiting, and pain.
* The first 10-minute part of the CD audio recordings prepared by the Turkish Psychologists Association is about deep relaxation.

purpose; The second 30-minute part includes instructions for relaxation exercises; The last 30 minutes are just it consists of relaxation music.

- In addition to standard treatment and care for laparoscopic cholecystectomy, volunteers who accept the study Progressive relaxation exercises were applied by the researcher at the 2nd, 6th, 12th and 24th hours after surgery.

When the literature review on PGE was made, it was seen that the application time and frequency of these exercises were not standard; 6th, 12th, 24th hours after surgery; It was applied on the 2nd day after surgery and the total number of sessions varied.

It is seen to show . In our study, PGE was detected at the 2nd, 6th, 12th and 24th hours after surgery.

has been implemented.Control group patients were informed about the research and received Informed Voluntary Consent Form (ANNEX-I) verbal and written permissions were obtained. - Before the surgery, the Patient Introduction Form (Annex-II) was checked both from the file and received verbal confirmation from the patient.

was filled in.

* The researcher was informed about the surgical intervention, expected nausea and vomiting, and pain.
* Patients in the control group were given the standard procedure for laparoscopic cholecystectomy only during the research period.

treatment and care were applied.

- No postoperative intervention was performed on the control group, and the researcher did not perform surgery after surgery.

Visual Comparison Scale (ANNEX-III) form for the severity of pain, nausea and vomiting at the 2nd, 6th, 12th and 24th hours The patient is asked to mark it with a pen or verbally indicate the severity between 1 and 10 on the form.

marking has been made.

* After the postoperative pain, nausea and vomiting status is determined on the Visual Comparison Scale, perioperative Patient Follow-up Form (ANNEX-IV) has been filled out.
* Data collection process of the research in order to eliminate ethical problems that may occur in the control group After completion, these patients were trained in progressive relaxation exercises.

ELIGIBILITY:
Inclusion Criteria:

* *To participate in the research willing

  * Prevents exercise creating a chronic without disease (COPD, heart failure etc.)
  * Hearing problem not found
  * At least primary school graduate the one which...
  * A psychiatric diagnosis non-major depression, anxiety disorders etc.) and anxiety or a drug for depression non-user
  * Elective laparoscopic having a cholecystectomy
  * Oriented to person, place and time the one which...
  * American Anesthesia Association(ASA) classification I, II or III the one which...

Exclusion Criteria:

Under 18 and over 70 patients over (n=2)

* Agree to participate in the research not (n=12)
* Patients undergoing emergency surgery
* Prevents exercise with disease causing
* Hearing problem found
* Having a psychiatric diagnosis (major depression, anxiety disorders etc.) and anxiety or a depression taking medication
* Pregnant
* Suffering from motion sickness
* Lack of cooperation
* Basic during surgery in life functions developing complications
* Open cholecystectomy (n=2)
* American Society of Anesthesiologists (ASA) classification IV are(n=7)
* Previous PGE exercises educated

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-08-25 (Actual)

PRIMARY OUTCOMES:
pain, nausea and vomiting 1 | at the 2nd hour after surgery
  The severity of pain, nausea, and vomiting was assessed by the researcher at the 2nd hour using a visual analog scale.

SECONDARY OUTCOMES:
pain, nausea and vomiting 2 | at the 6nd hours after surgery
  he severity of pain, nausea, and vomiting was assessed by the researcher at the 6th hour using a visual analog scale. vomiting at the 6th hours after surgery.
pain, nausea and vomiting 3 | at the 12th hour after surgery
  The severity of pain, nausea, and vomiting was assessed by the researcher at the 12 thhour using a visual analog scale.
pain, nausea and vomiting 4 | at the 24th hour after surgery
  The severity of pain, nausea, and vomiting was assessed by the researcher at the 24th hour using a visual analog scale.

CONTACTS AND LOCATIONS:
Overall Officials: Didem LAFÇI, associate professor, Study Director — Mersin University
Locations (1):
- Osmaniye State Hospital, Merkez, Osmani̇ye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
no ipd